CLINICAL TRIAL: NCT00240396
Title: Bimodal Analgesia as Form of Pain Control Post Long Bone Fracture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to enroll patients.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lars Richardson, Instructor in Orthopedic Surgery, Part-time, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005P000205
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Tibia Fracture; Femur Fracture; Humerus Fracture
Keywords: fracture; Tibia; femur; humerus; narcotics; bimodal; analgesia; long-bone; NSAIDS
MeSH Terms: conditions — Tibial Fractures; Femoral Fractures; Humeral Fractures; Fractures, Bone; Agnosia | interventions — Narcotics; Anti-Inflammatory Agents, Non-Steroidal

INTERVENTIONS:
Drug: Narcotics alone
Drug: Narcotics and NSAIDS

SUMMARY:
The purpose of this prospective randomized study is to evaluate the risks and benefits of using bimodal analgesia, (i.e. Narcotics and NSAIDS) vs Narcotics alone post long bone fracture.

DETAILED DESCRIPTION:
This will be a prospective, randomized, control trial looking at the benefit of bimodal analgesia in the treatment of long bone fractures. The traditional pain control regimen following fracture fixation typically involves a course of narcotics on an as-needed basis for pain relief. Recent data has shown that adding NSAIDS to the pain regimen as part of a bimodal approach to pain control, improves the efficacy of pain management and reduces narcotic use. Laboratory research on NSAIDs as it pertains to bone healing, however, has shown in animal models that there may be a positive association between NSAIDS and non-union rates. In other words, NSAIDS may prevent or delay bone healing. These results, however, have not been tested prospectively in humans.

The purpose of this study is to look at the combination of NSAIDS and narcotics post long bone fracture and monitor the effects on narcotic use and healing rates to ultimately and conclusively establish the risk or benefit of NSAIDS after long bone fracture.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patients over the age of 18 years
* Fracture of Tibia, femur, or Humerus.

Exclusion Criteria:

* Open fractures grade III
* Open fractures with suspected compartment syndrome
* history of prior fracture in particular limb.
* Concurrent usage of Steroid drugs, and immunosuppressants.
* Prior or current history of GI bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09-24 (Actual); Study Completion 2007-09-24 (Actual)

PRIMARY OUTCOMES:
pain score
Amount of narcotics used
time to fracture healing

SECONDARY OUTCOMES:
return to activity
complications
reoperation rate

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Richardson, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumont AS, Verma S, Dumont RJ, Hurlbert RJ. Nonsteroidal anti-inflammatory drugs and bone metabolism in spinal fusion surgery: a pharmacological quandary. J Pharmacol Toxicol Methods. 2000 Jan-Feb;43(1):31-9. doi: 10.1016/s1056-8719(00)00077-0. PMID 11091128
- [Background] Aspenberg P. Avoid cox inhibitors after skeletal surgery! Acta Orthop Scand. 2002 Oct;73(5):489-90. doi: 10.1080/000164702321022730. No abstract available. PMID 12440488
- [Background] Allami MK, Giannoudis PV. Cox inhibitors and bone healing. Acta Orthop Scand. 2003 Dec;74(6):771-2. doi: 10.1080/00016470310018351. No abstract available. PMID 14763714
- [Background] Brown KM, Saunders MM, Kirsch T, Donahue HJ, Reid JS. Effect of COX-2-specific inhibition on fracture-healing in the rat femur. J Bone Joint Surg Am. 2004 Jan;86(1):116-23. doi: 10.2106/00004623-200401000-00017. PMID 14711953
- [Background] Giannoudis PV, MacDonald DA, Matthews SJ, Smith RM, Furlong AJ, De Boer P. Nonunion of the femoral diaphysis. The influence of reaming and non-steroidal anti-inflammatory drugs. J Bone Joint Surg Br. 2000 Jul;82(5):655-8. doi: 10.1302/0301-620x.82b5.9899. PMID 10963160